CLINICAL TRIAL: NCT01838083
Title: A Double-blind, Randomized, Two-treatment Crossover Bioequivalence Study Comparing Two New Insulin Glargine Formulations Using the Euglycemic Clamp Technique in Subjects With Type 1 Diabetes Mellitus
Brief Title: Euglycemic Clamp Study Comparing Two New Insulin Glargine Formulations in Subjects With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PKD13560; 2012-005777-31 (EudraCT Number); U1111-1139-3755 (Other: UTN)
Record Dates: First submitted 2013-04-16; First posted 2013-04-23 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Type1 Diabetes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin glargine new formulation (test T formulation) (Experimental): Once daily for 6 days
  Interventions: Drug: Insulin glargine new formulation HOE901
- Insulin glargine new formulation (reference R formulation) (Experimental): Once daily for 6 days
  Interventions: Drug: Insulin glargine new formulation HOE901

INTERVENTIONS:
Drug: Insulin glargine new formulation HOE901 — Pharmaceutical form: solution Route of administration: subcutaneous

SUMMARY:
Primary Objective:

To demonstrate equivalence in exposure to insulin glargine given as test formulation T and reference formulation R in steady state conditions after 6 once-daily subcutaneous (SC) doses

Secondary Objective:

* To assess relative Pharmacodynamic activity of the insulin glargine test formulation T to the insulin glargine reference formulation R in steady state conditions after 6 once-daily SC doses
* To assess the safety and tolerability of the test and reference formulations of two new insulin glargine formulations

DETAILED DESCRIPTION:
Total study duration per subject: 29 to 64 days including screening visit

Duration of each part of the study for one subject:

* Screening: 3 to 21 days before 1st dosing (Day -21 to Day -3)
* Treatment Period 1 and 2: 8 days (dosing on 6 days)
* Washout between last/1st dosing days of the treatment periods: 7-21 days (preferentially 7 days) End-of-Study Visit: 7-10 days after last dosing

ELIGIBILITY:
Inclusion criteria :

* Male or female subjects, between 18 and 64 years of age, inclusive, with diabetes mellitus type 1 for more than one year
* Total insulin dose of < 1.2 U/kg/day
* Minimum usual basal insulin dose ≥ 0.2 U/kg/day
* Body weight between 50.0 kg and 110.0 kg, Body Mass Index between 18.5 and 30.0 kg/m2 inclusive
* Fasting negative serum C-peptide (< 0.3 nmol/L)
* Glycohemoglobin (HbA1c) ≤ 75 mmol/mol [≤ 9.0%]
* Stable insulin regimen for at least 2 months prior to inclusion in study
* Certified as otherwise healthy for Type-1 Diabetes mellitus patient
* Laboratory parameters within the normal range
* Women of childbearing potential with negative pregnancy test and use of a highly effective contraceptive method or women with confirmed postmenopausal status

Exclusion criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic (apart from diabetes mellitus type 1), hematological, neurological, psychiatric, systemic (affecting the body as a whole), ocular, gynecologic (if female), or infectious disease; any acute infectious disease or signs of acute illness.
* More than one episode of severe hypoglycemia with seizure, coma or requiring assistance of another person during the past 6 months
* Frequent severe headaches and / or migraine, recurrent nausea and / or vomiting (more than twice a month)
* Symptomatic hypotension (whatever the decrease in blood pressure), or asymptomatic postural hypotension defined by a decrease in systolic blood pressure equal to or greater than 20 mmHg within three minutes when changing from the supine to the standing position
* Presence or history of a drug allergy or clinically significant allergic disease according to the Investigator's judgment
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol
* Presence or history of drug or alcohol abuse (alcohol consumption > 40 grams / day)
* If female, pregnancy (defined as positive Beta Human Chorionic Gonadotropin test), breast-feeding
* Known hypersensitivity to insulin glargine or excipients of the study drug
* Any history or presence of deep leg vein thrombosis or a frequent appearance of deep leg vein thrombosis in first degree relatives (parents, siblings or children)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin concentration curve within 24 hours (INS-AUC0-24) after dosing on Day 6 | 24-hours (D6 to D7)

SECONDARY OUTCOMES:
Maximum insulin concentration (INS-Cmax) | 24-hours (D6 to D7)
Time to INS-Cmax (INS-tmax) | 24-hours (D6 to D7)
Time to reach 50% of INS-AUC0-24 (T50%-INS-AUC0-24) | 24-hours (D6 to D7)
Area under the body-weight-standardized Glucose Infusion Rate (GIR) within 24 hours (GIR-AUC0-24h) after dosing on Day 6 during the clamp | 24-hours (D6 to D7)
Maximum smoothed body weight standardized glucose infusion rate (GIRmax) | 24-hours (D6 to D7)
Time to GIRmax (GIR-Tmax) | 24-hours (D6 to D7)
Time to reach at least 50% of GIR-AUC0-24 (T50%-GIR-AUC0-24) | 24-hours (D6 to D7)
Duration of blood glucose control (time to elevation of smoothed blood glucose profile above clamp level and to elevation above different prespecified blood glucose levels) | 24-hours (D6 to D7)
Safety as measured by adverse events/serious adverse events, ohypoglycemia events, physical examinations, clinical laboratory, electrocardiograms, vital signs, injection site reactions and anti-insulin antibodies. | up to 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 276001, Neuss, Germany